CLINICAL TRIAL: NCT07143734
Title: A Pilot Randomized Placebo-Controlled Trial of Transcranial Pulse Stimulation (TPS) in Early Alzheimer's Disease (AD) Subjects
Brief Title: Transcranial Pulse Stimulation for Alzheimer's Disease
Acronym: TPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Asia Pacific Institute of Healthy ageing (Unknown); Associated medical supplies company limited (Unknown); Dongguan University of Technology (Unknown); SuZhou Engin Bio-medical Electronics.Co.Ltd. (Unknown)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024.645
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Dementia (AD)
Keywords: Transcranial Pulse Stimulation (TPS); Alzheimer Dementia (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants with early AD, confirmed via blood tests, are randomly assigned to either a TPS treatment group or a placebo group. The treatment protocol involves an intensive TPS treatment period over two weeks followed by a continuous treatment period with additional treatments over some weeks. The placebo group receives sham treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Received transcranial pulse stimulation (TPS) treatment (Experimental): Receiving transcranial pulse stimulation (TPS) as part of an investigation into its effectiveness for improving cognitive function, memory, functional status, and neuropsychiatric symptoms in subjects with Alzheimer's Disease (AD).
  Interventions: Device: transcranial pulse stimulation (TPS)
- Received transcranial pulse stimulation (TPS) sham treatment (Sham Comparator): Participants will undergo an identical procedure using a device that mimics the sound and sensation of active TPS but delivers no therapeutic energy pulses to the brain.
  Interventions: Device: transcranial pulse stimulation (TPS-Sham)

INTERVENTIONS:
Device: transcranial pulse stimulation (TPS) — The TPS/Sham-TPS therapy is administered for the first two weeks, followed by additional sessions at some week intervals.
  Arms: Received transcranial pulse stimulation (TPS) treatment
Device: transcranial pulse stimulation (TPS-Sham) — Participants will undergo an identical procedure using a device that mimics the sound and sensation of active TPS but delivers no therapeutic energy pulses to the brain.
  Arms: Received transcranial pulse stimulation (TPS) sham treatment

SUMMARY:
TPS is a non-invasive therapeutic modality that uses focused, low-energy pulse stimulation to stimulate tissue regeneration and reduce inflammation. In the context of neurological disorders, it is hypothesized that TPS can modulate neuronal activity, enhance synaptic plasticity, and reduce neuroinflammation. It is a relatively new application in neurological disease treatment and is still under intense investigation.

DETAILED DESCRIPTION:
This pilot randomized placebo-controlled trial investigates the effects of transcranial pulse stimulation in subjects with early Alzheimer's Disease (AD). The TPS/Sham-TPS is administered for the first two weeks, followed by additional sessions at some week intervals. The transcranial pulse stimulation device used in this trial is a CE-certified medical instrument (ISO 9001 and ISO 13485).

The study aims to evaluate cognitive function, and neuropsychiatric symptoms using the some cognitive assessment tools, Frontal near-infrared spectroscopy (fNIRS), and fasting blood test at baseline at week 12.

This study is expected to lay the groundwork for future, larger-scale studies

ELIGIBILITY:
Inclusion Criteria:

* Adults who have been clinically diagnosed with Alzheimer's Disease in the early stage 2-6a according to the Functional Assessment Staging Test (In Appendix A)
* The mental capacity to give informed consent for research is made by an experienced geriatrician based on Appendix A.
* Aged 60-90 years old.
* Able to make informed consent under assistance, which is witnessed and signed by a family caregiver.

Exclusion Criteria:

* Cannot understand Chinese.
* Mentally incapacitated, unable to provide informed consent
* Inability to remain still for 30 minutes
* Lack of available family caregiver to answer questionnaires
* Alcohol or substance dependence
* Major neurological conditions, including:
* Brain tumor
* Brain aneurysm
* Presence of any metal implants in the brain
* Hemophilia or other blood clotting disorders
* History of thrombosis

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale score. | baseline（ 1st Week）； follow-up （ after finishing the TPS therapy at 12th week）
  The lower the score, the better the cognitive function; the higher the score, the more severe the cognitive impairment.
  Score range: 0-85

SECONDARY OUTCOMES:
Change in the Neuropsychiatric Inventory total score. | baseline（ 1st Week）； follow-up （ after finishing the TPS therapy at 12th week）
  The lower the score, the milder the neuropsychiatric symptoms; the higher the score, the more severe and frequent the symptoms, and the greater the burden on caregivers.
  Score range： 0-144
Change in the Animal Fluency Test score | baseline（ 1st Week）； follow-up （ after finishing the TPS therapy at 12th week）
  The more animal names you say within the specified time (the higher the score), the better your language fluency, cognitive processing speed, and semantic memory ability.
  Normal cognition typically has ≥ 15-18 (well-educated young or middle-aged individuals typically have ≥ 20).
  Mild cognitive impairment (MCI) may have 11-16 Dementia (such as Alzheimer's disease) typically has ≤ 12-14 , but may be lower.
Change in the Disability Assessment for Dementia total score. | baseline（ 1st Week）； follow-up （ after finishing the TPS therapy at 12th week）
  The higher the score, the greater the patient's functional independence and the better the ability to carry out daily life. The lower the score, the more severe the functional impairment and the greater the dependence on others for care.
  Score range：0-100%
Change in oxygenated hemoglobin (HbO) and deoxygenated hemoglobin (HbR) in the cerebral blood | baseline（ 1st Week）； follow-up （ after finishing the TPS therapy at 12th week）
Change in plasma Aβ42/40 | baseline（ 1st Week）； follow-up （ after finishing the TPS therapy at 12th week）

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Chi Yui Kwok, PhD, Principal Investigator — Department of Medicine & Therapeutics, Faculty of Medicine, The Chinese UNiversity of Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Faculty of Medicine, The Chinese UNiversity of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This is official website of the Neurolith Transcranial Pulse Stimulation device — https://www.storzmedical.com/en/disciplines/tps-products-for-the-treatment-of-alzheimer-s-disease/neurolith/